CLINICAL TRIAL: NCT00387166
Title: Cardiovascular Risk Disparities: Socio-Emotional Pathways
Brief Title: Socioeconomic Status, Psychosocial Factors, and CVD Risk in Mexican-American Women
Status: Completed | Type: Observational
Sponsor: San Diego State University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Linda C. Gallo, Professor, San Diego State University
Other Study IDs: 1339; R01HL081604-01A1 (NIH); G00006532
Record Dates: First submitted 2006-10-11; First posted 2006-10-12 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: Hypertension; Cardiovascular Disease; Metabolic Disorders
Keywords: Type 2 Diabetes; Cardiovascular; Blood Pressure; Hispanic; Women; Social Context; Psychosocial
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases; Metabolic Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine specimens were collected to identify stress hormones and inflammatory markers. Whole blood, plasma, and serum are stored for possible future assays based on new discoveries.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: Mexican-American women, aged 40-65

SUMMARY:
Cardiovascular disease (CVD) is the leading cause of death in American women, claiming on average 40% of all female deaths each year. Although the number of CVD-related deaths in the United States has decreased over the last several decades, the rate of decline has been less for women than for men. Specifically, minority women of low socioeconomic status make up a disproportionately high number of CVD cases and related deaths. Previous studies suggest that, in addition to many other variables, psychosocial variables may contribute to ethnic CVD disparities. More research, however, is needed to help understand and reduce these differences. This study will examine the associations among socioeconomic status, psychological and social factors, CVD biomarkers, and CVD in Mexican-American women.

DETAILED DESCRIPTION:
One in four women in the United States has some form of CVD, which includes heart disease, high blood pressure, and heart attack. Minority and low socioeconomic status populations show particularly disproportionate rates of CVD morbidity and mortality. Previous research suggests that individuals with lower social status may suffer negative emotional and physical health consequences due to increased stress experienced across multiple areas of life. It is believed that stress may directly affect behavioral, physiological, and emotional risk processes, which have all been linked to increased CVD risk. In addition, people with low socioeconomic status are often less capable of seeking psychosocial resources with which to manage stress, making them especially vulnerable to the associated physical and emotional wear and tear. More information is needed on the effects of psychosocial variables on the cardiovascular health of minority, specifically Mexican-American, women. This study will examine the associations among socioeconomic status, psychological and social factors, CVD biomarkers, and CVD in Mexican-American women.

Participation in this study will involve two home visits, with total participation time lasting about 6 hours. During the first study visit, participants will complete a variety of questionnaires on stressful experiences, social relationships, background and culture, thoughts and emotions, health habits, and medical history. Participants will also have their blood pressure measured and will be given a container and instructions to perform a 12-hour overnight urine collection.

During the second study visit, occurring a couple of days after the first visit, participants will undergo a blood draw, physical and vital sign measurements, and a training session on how to use an ambulatory blood pressure monitor and handheld computer diary. Participants who fit properly into the arm cuff of the ambulatory blood pressure monitor will then be asked to wear the monitor for 36 hours. Every time the monitor records a blood pressure reading, participants will be asked to use their handheld computer diary and answer questions about temperature, exercise, posture, stress, mood, and social interactions. There will be a total of 52 to 56 diary entries, taking between 2 and 3 minutes to complete each entry. Within 1 month, participants will receive a letter summarizing their health profile in terms of weight, cholesterol levels, and blood glucose. Participants will also be provided with information on seeking appropriate treatments for any health problems discovered on their profile.

ELIGIBILITY:
Inclusion Criteria:

* Self identifies as Mexican-American
* Resides in Chula Vista or National City
* Sufficiently mobile to complete ambulatory blood pressure assessment

Exclusion Criteria:

* Pregnant
* Current or historical cardiovascular disease
* Current Type II diabetes
* Cancer treatment in the 10 years before study entry
* Bleeding disorder
* Use of medications with autonomic effects

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include healthy Mexican-American women from the South San Diego community.
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 2006-10; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Stress, psychosocial risk and resilient factors, socio-cultural factors, and bio-behavioral markers of cardiovascular risk | Measured at completion of sample analysis

CONTACTS AND LOCATIONS:
Overall Officials: Linda C. Gallo, PhD, Principal Investigator — San Diego State University; John Elder, PhD, Principal Investigator — San Diego State University; Paul Mills, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- San Diego State University, Institute for Behavioral and Community Health, San Diego, California, United States

REFERENCES:
- [Background] Gallo LC, Matthews KA. Understanding the association between socioeconomic status and physical health: do negative emotions play a role? Psychol Bull. 2003 Jan;129(1):10-51. doi: 10.1037/0033-2909.129.1.10. PMID 12555793
- [Background] Matthews KA, Gallo LC. Psychological perspectives on pathways linking socioeconomic status and physical health. Annu Rev Psychol. 2011;62:501-30. doi: 10.1146/annurev.psych.031809.130711. PMID 20636127
- [Background] Gallo LC, Penedo FJ, Espinosa de los Monteros K, Arguelles W. Resiliency in the face of disadvantage: do Hispanic cultural characteristics protect health outcomes? J Pers. 2009 Dec;77(6):1707-46. doi: 10.1111/j.1467-6494.2009.00598.x. Epub 2009 Sep 30. PMID 19796063
- [Result] Gallo LC, Fortmann AL, Roesch SC, Barrett-Connor E, Elder JP, de los Monteros KE, Shivpuri S, Mills PJ, Talavera GA, Matthews KA. Socioeconomic status, psychosocial resources and risk, and cardiometabolic risk in Mexican-American women. Health Psychol. 2012 May;31(3):334-42. doi: 10.1037/a0025689. Epub 2011 Nov 7. PMID 22059620
- [Result] Gallo LC, Jimenez JA, Shivpuri S, Espinosa de los Monteros K, Mills PJ. Domains of chronic stress, lifestyle factors, and allostatic load in middle-aged Mexican-American women. Ann Behav Med. 2011 Feb;41(1):21-31. doi: 10.1007/s12160-010-9233-1. PMID 20878511
- [Result] Gonzalez P, Castaneda SF, Mills PJ, Talavera GA, Elder JP, Gallo LC. Determinants of breast, cervical and colorectal cancer screening adherence in Mexican-American women. J Community Health. 2012 Apr;37(2):421-33. doi: 10.1007/s10900-011-9459-2. PMID 21874364
- [Result] Shivpuri S, Gallo LC, Mills PJ, Matthews KA, Elder JP, Talavera GA. Trait anger, cynical hostility and inflammation in Latinas: variations by anger type? Brain Behav Immun. 2011 Aug;25(6):1256-63. doi: 10.1016/j.bbi.2011.04.016. Epub 2011 May 1. PMID 21554946
- [Derived] Gallo LC, Fortmann AL, de Los Monteros KE, Mills PJ, Barrett-Connor E, Roesch SC, Matthews KA. Individual and neighborhood socioeconomic status and inflammation in Mexican American women: what is the role of obesity? Psychosom Med. 2012 Jun;74(5):535-42. doi: 10.1097/PSY.0b013e31824f5f6d. Epub 2012 May 11. PMID 22582313
- See also: More information at the Institute for Behavioral and Community Health (IBACH) Webpage — http://www.ibachsd.org/